CLINICAL TRIAL: NCT03200197
Title: Effectiveness of Menthol Chewing Gum in the Management of Preoperative Thirst: Randomized Clinical Trial
Brief Title: Effectiveness of Menthol Chewing Gum in the Management of Thirst
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Estadual de Londrina (Other)
Responsible Party: Principal Investigator, Aline Korki Arrabal Garcia, Master of Science Degree in Nursing, Universidade Estadual de Londrina
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Aline Korki Arrabal Garcia
Record Dates: First submitted 2017-06-22; First posted 2017-06-27 (Actual); Last update posted 2017-06-27 (Actual); Status verified 2017-06

CONDITIONS: Thirst
Keywords: Chewing gum; Artificial saliva; Saliva; Mastication; Salivary glands; Xerostomia
MeSH Terms: conditions — Xerostomia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- menthol chewing gum (Experimental): Allocation concealment was performed through the use of individual opaque envelopes numbered externally in sequence, containing the randomly defined group information.This step was performed by a researcher who did not participate in the data collection. The intensity of the initial thirst was measured by means of the Verbal Numerical Scale (VNS), which ranged from 0 (no thirst) to 10 (very intense thirst) and the discomfort of the initial thirst was measured through the Perioperative Thirst Discomfort Scale (PTDS), which is composed of 7 attributes and ranges from 0 to 14. After using the intervention (menthol chewing gum) for 10 minutes, chewing at a natural rhythm and swallowing the saliva produced, the intensity and final discomfort were measured using the same scales.
  Interventions: Other: Menthol chewing gum
- Usual care (maintenance of fasting) (Active Comparator): Allocation concealment was performed through the use of individual opaque envelopes numbered externally in sequence, containing the randomly defined group information.This step was performed by a researcher who did not participate in the data collection.The intensity of the initial thirst was measured by means of the Verbal Numerical Scale (VNS), which ranged from 0 (no thirst) to 10 (very intense thirst) and the discomfort of the initial thirst was measured through the Perioperative Thirst Discomfort Scale (PTDS), which is composed of 7 attributes and ranges from 0 to 14. After maintaining the usual care, that is, reaffirming the need for fasting for 10 minutes, the intensity and final discomfort were measured using the same scales.
  Interventions: Other: Usual care (fasting)

INTERVENTIONS:
Other: Menthol chewing gum — The experimental group received one unit of mentholated chewing gum, chewing and swallowing the saliva in a natural rhythm for 10 minutes. The menthol chewing gum used is called TRÍDENT®and is composed as follows: base gum, hydrogenated vegetable oil, vegetable oil, sweeteners: sorbitol, xylitol, mannitol, maltitol, aspartame, acesulfame potassium, and sucralose, humectants: glycerin and triacetin, flavorings (contains wheat derivatives), anti-humectant talc, emulsifiers: esters of mono- and diglycerides of fatty acids with acetic acid, soy lectin and mono and diglycerides of fatty acids and colorings: tartrazine and brilliant blue FCF, presenting a weight of 1.8g per unit.
  Arms: menthol chewing gum
Other: Usual care (fasting) — The control group received the usual care given at the hospitalization units, that is, when the patient reported thirst, the need to maintain fasting for 10 minutes was reaffirmed.
  Arms: Usual care (maintenance of fasting)

SUMMARY:
The objective of this study was to compare the effectiveness of menthol chewing gum compared to maintained fasting (usual care) in reducing the intensity of the surgical patient's thirst during the preoperative period. The hypothesis of the study was that the use of menthol chewing gum in surgical patients in the preoperative period would be more effective than the maintenance of fasting with regard to the decrease in thirst and its discomforts.

DETAILED DESCRIPTION:
There is evidence that chewing gum is effective in relieving thirst in the surgical patient in the preoperative period as it stimulates the salivary glands by means of mechano and chemoreceptors, increasing the salivary pH and flow, lubricating the oral cavity, acting in this way on peripheral thirst, which is triggered by dehydration of the oral mucosa. Furthermore, menthol gum stimulates the cold receptors, known as TRPM8, which are responsible for deactivating centers of thirst. Thus, the risk of bronchoaspiration due to gastric fullness is avoided and the discomfort of a dry mouth is reduced.Preliminary evidence indicates that the chewing gum strategy assists in the relief of a dry mouth and thirst in patients undergoing dialysis and head and neck radiotherapy. However, there is no scientific evidence of controlled studies with results that can be generalized regarding the use of chewing gum to reduce thirst and its discomforts in surgical patients in the preoperative period when they remain in a fasted state.

ELIGIBILITY:
Inclusion Criteria:

* Elective Surgeries;
* Aged between 12 and 65 years;
* Did not receive preanesthetic medication;
* Oriented in time and space;
* Present dentition (natural or artificial);
* Fasting for a minimum of three hours;
* Available for collection at least 3 hours prior to the scheduled surgical procedure;
* Verbalize thirst spontaneously or when questioned with an intensity greater than or equal to three on the Verbal Numerical Scale (VNS);

Exclusion Criteria:

* Allergy to menthol;
* Chewing restriction;
* Swallowing restriction;
* Patients who presented nausea, vomiting, or pain;
* Patients with chronic xerostomia;
* Chronic renal patients;

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
intensity of thirst | 10 minutes
  Alteration in the evaluation of the final intensity of thirst in relation to the evaluation of the initial intensity of thirst [10 minutes]. For evaluation of the intensity of thirst, a Verbal Numeral Scale (VNS) was used, with a range from 0 (no thirst) to 10 (very intense thirst), as reported by the patients when questioned.

SECONDARY OUTCOMES:
discomfort of thirst | 10 minutes
  Alteration in the evaluation of the final discomfort of thirst in relation to the evaluation of the initial discomfort of thirst [10 minutes]. The Perioperative Thirst Discomfort Scale (PTDS) was used to evaluate the discomfort of the thirst.This scale is composed of 7 attributes that evaluate the signs of discomfort of perioperative thirst, as follows: dry mouth, dry lips, thick tongue, thick saliva, bad taste in the mouth, and desire to drink water. Each attribute varies between 0 (no inconvenience), 1 (a little inconvenient), and 2 (very inconvenient). The final sum of the PTDS can range from 0 to 14 points.

CONTACTS AND LOCATIONS:
Overall Officials: Ligia Fahl Fonseca, Study Director — State University of Londrina

IPD SHARING:
Plan to Share IPD: Undecided